CLINICAL TRIAL: NCT01344694
Title: Association Between Epicardial Fat, Visceral Fat Accumulation & Cardiovascular Atherosclerosis
Brief Title: Epicardial Fat, Visceral Fat and Coronary Atherosclerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Dr. Assy Nimer, Ziv Medical center
Other Study IDs: 0020-11
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-04

CONDITIONS: Epicardial Fat; Visceral Fat; Atherosclerosis
Keywords: Epicardial fat; Visceral fat; atherosclerosis; coronary computed tomography angiography; Carotid Doppler ultrasound
MeSH Terms: conditions — Atherosclerosis | interventions — 6-pyruvoyltetrahydropterin synthase

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- patient with liver fat: 30 patients with liver fat
  Interventions: Other: patient with liver fat
- excess of visceral fat: 50 pts. with excess of visceral fat
  Interventions: Other: pts. with excess of visceral fat
- control: 30 control subjects
  Interventions: Other: control

INTERVENTIONS:
Other: patient with liver fat — 30 patient with liver fat
  Groups: patient with liver fat
Other: pts. with excess of visceral fat — pts. with excess of visceral fat
  Groups: excess of visceral fat
Other: control — 30 control subjects
  Groups: control

SUMMARY:
Background: Visceral fat is increasingly associated with metabolic syndrome and with fatty liver, a condition carrying a high risk of cardiovascular disease. The independent role of epicardial fat deposition in cardiovascular risk remains unclear.

DETAILED DESCRIPTION:
Background: Visceral fat is increasingly associated with metabolic syndrome and with fatty liver, a condition carrying a high risk of cardiovascular disease. The independent role of epicardial fat deposition in cardiovascular risk remains unclear. Aim: Evaluate the link between epicardial fat, visceral fat, liver fat accumulation and cardiovascular diseases and carotis atherosclerosis in patients with the major cardiovascular risk factors and with or without metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to cardiac CT will be the source of recruitment.
* patients with excess of visceral fat,
* 30 patients with liver fat accumulation
* 30 sex-age-matched individual (controls) will be enrolled. All patients will undergo a complete family history, personal clinical history, physical examination and blood sampling for biochemical analysis.
* Informed consent will be obtained from each individual.

Exclusion Criteria:

* subjects with severe morbid obesity (body mass index [BMI] > 40),
* recent history of acute illness,
* clinical history of ischemic heart disease and cerebrovascular disease,
* typical chest pain,
* previous coronary artery disease,
* conventional coronary angiography, percutaneous interventions, coronary by pass grafting, renal failure, cancer patients,
* subjects who take drugs that induces hepatic steatosis ( corticosteroids, estrogens, methotrexate, amiodarone and others)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 patients (age 40-70) with excess of visceral fat (obese), 30 patient with liver fat and 30 sexes, age matched individuals will be recruited.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-02 (Estimated); Study Completion 2012-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nimer Assy, md, Principal Investigator — Ziv MC
Locations (1):
- Ziv MC, Safed, Israel